CLINICAL TRIAL: NCT01314365
Title: DYSPORT™ for Injection AbobotulinumtoxinA Neurotoxin Clinical & Health Economics Outcomes Registry in Cervical Dystonia (ANCHOR-CD)
Brief Title: DYSPORT™ Clinical & Health Economics Outcomes Registry in Cervical Dystonia
Acronym: ANCHOR-CD
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-TL-52120-156
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the protocol is to determine typical patient response to Dysport in the treatment of adult cervical dystonia (CD).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic CD as determined by the enrolling investigator
* If previously treated with a neurotoxin for CD, at least a 12-week interval must have elapsed between the last injection of Botulinum toxin A (BoNT-A) or Botulinum toxin B (BoNT-B) and the first dose of Dysport injected in this study
* Patient is able to comply with the protocol (e.g., can visit the clinic as required and can complete questionnaires/telephone interviews)
* Provision of written informed consent prior to enrollment

Exclusion Criteria:

* Contraindications to treatment with any BoNT-A or BoNT-B preparations
* Based on Investigator opinion, patients in whom previous BoNT-A or BoNT-B therapy has failed to produce a clinical response or produced an intolerable adverse reaction
* Anticipated concomitant treatment with BoNT for other than cervical dystonia
* Secondary cervical dystonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Cervical Dystonia treated with Dysport
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of treatment responders using the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) severity scale score | Cycle 1 - Baseline and week 4
Patient Global Impression of Change using the 7-point Likert scale | Cycle 1 - Baseline and week 4

SECONDARY OUTCOMES:
Clinical Global Impression of Change using the 7-point Likert scale | Cycle 1 - Week 4 and early termination visit
Patient Global Impression of Change using the 7-point Likert scale | Cycle 1 - Week 4; Cycles 2 to 4 - Baseline, week 4 and termination visits
Time to Waning Effect of Dysport treatment/symptom re-emergence | Cycles 1 to 4 - Week 8 and at study termination visits
Patient-self-administered questionnaire (Cervical Dystonia Impact Profile-58) | Cycles 1 & 3: Baseline
Patient-reported assessment of pain using the Pain Numeric Rating Scale (NRS) | Cycles 1 to 4 - Baseline, week 4 and at study termination visits
Treatment Satisfaction Questionnaire for Medication (TSQM) | Cycle 1 - Week 4; Cycles 2 to 4 - Baseline, week 4 and termination visit

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (45):
- United States (45):
  - Arizona Dystonia Institute, Scottsdale, Arizona
  - East Bay Physicians Medical Group, Berkeley, California
  - Headache Center, Encinitas, California
  - The Parkinson's & Movement Disorder Institute, Fountain Valley, California
  - Neuro-Pain Medical Center, Fresno, California
  - Coastal Neurological Medical Group, Inc., La Jolla, California
  - Valley Parkinson Clinic, Los Gatos, California
  - Harvinder S. Birk, Redding, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - University of Colorado Denver, Denver, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - University of Miami, Dept. of Movement Disorders Clinic, Miami, Florida
  - Palm Beach Gardens Medical Center, North Palm Beach, Florida
  - Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - Parkinson's Treatment Center of SW Florida, Port Charlotte, Florida
  - USF HealthParkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Elks Rehab Hospital - Movement Disorders Center, Boise, Idaho
  - Rush University Medical Center Department of Neurological Sciences, Chicago, Illinois
  - Kansas City Bone & Joint Clinic, PA Overland Park, Overland Park, Kansas
  - Baptist Neurology Center - Lexington, Lexington, Kentucky
  - The Neuro Medical Center, Baton Rouge, Louisiana
  - The Parkinson's and Movement Disorders Center, Southfield, Michigan
  - Rehabilitation Consultants, PA, Eagan, Minnesota
  - Methodist Rehabilitation Center, Jackson, Mississippi
  - University of Nevada School of Medicine, Reno, Nevada
  - Empire Neurology PC, the MS Center of Northeastern New York, Latham, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Riverhills Neuroscience, Cincinnati, Ohio
  - University Neurology, Inc., Cincinnati, Ohio
  - Cleveland Clinic Center for Neurological Restoration, Cleveland, Ohio
  - Capital Neurology Services & MS Institute, Gahanna, Ohio
  - Neurological Associates of Tulsa, Tulsa, Oklahoma
  - Columbia Pain Management, PC, Hood River, Oregon
  - Allegheny General Hospital_Department of Neurology, Pittsburgh, Pennsylvania
  - Coastal Neurology, PA, Port Royal, South Carolina
  - Victorium Clinical Research, San Antonio, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - Gershon Pain Specialists, Virginia Beach, Virginia
  - Evergreen Hospital Medical Center/Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - South Puget Sound Neurology, Tacoma, Washington
  - Gundersen Clinic, Ltd., La Crosse, Wisconsin

REFERENCES:
- [Derived] Trosch RM, Misra VP, Maisonobe P, Om S. Impact of abobotulinumtoxinA on the clinical features of cervical dystonia in routine practice. Clin Park Relat Disord. 2020 Jun 15;3:100063. doi: 10.1016/j.prdoa.2020.100063. eCollection 2020. PMID 34316644
- [Derived] Espay AJ, Trosch R, Suarez G, Johnson J, Marchese D, Comella C. Minimal clinically important change in the Toronto Western Spasmodic Torticollis Rating Scale. Parkinsonism Relat Disord. 2018 Jul;52:94-97. doi: 10.1016/j.parkreldis.2018.03.002. Epub 2018 Mar 7. PMID 29530726